CLINICAL TRIAL: NCT05051072
Title: Assessment in Patients With Essential Trigeminal Neuralgia of Nerve Involvement by MRI in DTI and Functional Connectivity in "Resting State"
Acronym: SENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLL_2020_37
Record Dates: First submitted 2021-09-09; First posted 2021-09-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Trigeminal Neuralgia; Microvascular Decompression Surgery; Diffusion Tensor Imaging
Keywords: Resting state
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI in morphological sequence, diffusion tensor and resting functional (Other): * standard anatomical sequences T1, FLAIR (Fluid Attenuated Inversion Recovery), TOF(Time-of-flight MR angiography) , DRIVE, sequence centered on the V after injection of gadolinated contrast product as part of routine care,
  * diffusion tensor sequence (DTI)
  Interventions: Procedure: Assessment of the trigeminal nerve by diffusion tensor MRI and in "resting state" in the context of essential neuralgia

INTERVENTIONS:
Procedure: Assessment of the trigeminal nerve by diffusion tensor MRI and in "resting state" in the context of essential neuralgia — Assessment of the trigeminal nerve by diffusion tensor MRI and in "resting state" in the context of essential neuralgia

SUMMARY:
Essential trigeminal neuralgia is the most common facial pain. In forms resistant to drug and disabling treatments, surgical treatment may be offered to the patient. The type of intervention will be conditioned by the presence or absence of a vasculo-nervous conflict objectified by MRI(Magnetic resonance imaging) Morphological MRI with contrast injection does not always allow an accurate assessment of trigeminal nerve damage in patients with essential facial neuralgia. Despite advances in the anatomical definition of high-resolution MRI, the correlation between a vascular conflict visible on MRI and present during surgery and prolonged postoperative clinical improvement remains insufficient These data raise the question of additional imaging sequences to assess the distressing characteristics of NT in addition to the usual anatomical criteria for compression By performing during morphological MRI two additional sequences, one in diffusion tensor (DTI) and one in resting state (fMRI), we could better characterize the achievement of NT

The contribution of new imaging sequences in the context of essential trigeminal neuralgia treated with microvascular decompression (MVD) would:

1/improve the diagnostic criteria for suffering and compression of the NT (trigeminal nerve) 2 / define objective prognostic criteria for the effectiveness of surgery, particularly in the context of unusual clinical symptoms or moderate conflict on MRI (Magnetic resonance imaging) 3 / to analyze more precisely the causes of recurrence at a distance from surgery and help in the decision of re-intervention Our main hypothesis: the addition of a diffusion tensor sequence and sequences (allowing functional brain analysis) in addition to standard anatomical MRI in the assessment of a vasculo-nervous conflict would allow us to better characterize involvement of the trigeminal nerve in essential facial neuralgia. It also helps guide therapeutic management and surgical indications.

This is a prospective, monocentric cohort study. It will be offered to patients referred to neurosurgery or to the pain assessment and treatment center for assessment and management of a neuralgia of the essential trijumeau unilateral.

DETAILED DESCRIPTION:
Name:

MRI in morphological sequence, diffusion tensor and resting functional

Description:

The MR exam will be performed on the Neuroradiology 3 Tesla (Philips) MR according to the following protocol:

* Standard anatomical sequences T1, FLAIR, TOF, DRIVE, sequence centered on the V after injection of gadolinated contrast product as part of standard care
* Diffusion tensor sequence (DTI) It allows the analysis of encephalic white matter beams in healthy subjects as well as in many pathologies
* resting state sequence (fMRI) This sequence is based on the spontaneous correlation of the BOLD signal (blood-oxygen level dependent) between different distant brain regions.
* The total duration of the exam will be about 45 minutes, including 15 minutes for the sequences added by the search.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and over);
* Supported in the neurosurgery department or at the assessment and treatment center for pain for unilateral essential trigeminal neuralgia with search for vasculo-nervous conflict;

Exclusion Criteria:

* Patient with neurodegenerative or inflammatory neurological pathology;
* Patient who has already been operated on for a DMV;
* Absolute contraindication to MRI
* Patient benefiting from a legal protection measure; with impaired judgment skills or unable to receive information;
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of micro-structural changes in the trigeminal nerve in essential neuralgia | Day 0 - inclusion
  Describe in patients with unilateral essential trigeminal neuralgia, the micro-structural modifications of the trigeminal nerve observed from data from the DTI sequence compared to the healthy contralateral side

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No